CLINICAL TRIAL: NCT06357572
Title: Real-life Clinical FEIBA Samples Measured Using the Version A of the HemA EnzySystem
Status: Completed | Type: Observational
Sponsor: Enzyre B.V. (Industry)
Collaborators: Instytut Hematologii i Transfuzjologii, Warschau, Poland (Unknown)
Responsible Party: Sponsor
Other Study IDs: ENZ13-2024
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Hemophilia A With Inhibitor; Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemophilia A patients prophylactically treated with FEIBA
  Interventions: Diagnostic Test: Thrombin generation assay (EnzySystem HemA version A - whole blood); Diagnostic Test: Thrombin generation assay (Ceveron s100 (Technoclone) - fresh plasma); Diagnostic Test: Additional coagulation tests

INTERVENTIONS:
Diagnostic Test: Thrombin generation assay (EnzySystem HemA version A - whole blood) — Whole blood obtained by venipuncture is immediately tested with the EnzySystem HemA version A), before and 0, 30, 120 and 240 minutes after administration of FEIBA.
Diagnostic Test: Thrombin generation assay (Ceveron s100 (Technoclone) - fresh plasma) — Whole blood is centrifuged to obtain plasma. The fresh plasma is tested using the Ceveron s100.
Diagnostic Test: Additional coagulation tests — Plasma samples are frozen for later coagulation testing. The following tests are performed:
  Factor VIII activity von Willebrand Factor antigen levels von Willebrand Factor ristocetin activity levels Prothrombin Fragment 1+2 levels ADAMTS13 activity FVIII antigen levels Nijmegen Hemostasis Assay

SUMMARY:
The goal of this observational study is to assess if the version A of the HemA EnzySystem, a novel portable coagulation testing platform, can be used in patients with hemophilia A treated with Factor VIII Bypassing Agent (FEIBA). The main question[s] it aims to answer are:

* Can the version A of the HemA EnzySystem can record thrombin generation within a time frame of 60 min in fresh whole blood samples of patients with hemophilia A treated with FEIBA?
* Are the TGA results of the version A of the HemA EnzySystem in agreement with the TGA results obtained with conventional methods in fresh non frozen plasma?

Participants are asked to fill in a questionnaire regarding their general health and hemophilia treatment. Subsequently, blood will be drawn from the patients before, and at 30, 120, and 240 minutes after FEIBA administration. Whole blood is immediately tested using the Version A HemA EnzySystem, and plasma is generated for testing with the Ceveron s100 (Technoclone). Leftover samples are frozen for later additional coagulation testing.

DETAILED DESCRIPTION:
Rationale: Hemophilia is an X-linked hemostatic bleeding disorder characterized by a lack of coagulation factor VIII activity (HemA) or factor IX activity (HemB). Spontaneous major bleeding in joints and muscles frequently occur when factor activity levels are low. Currently, there is a growing evidence that the bleeding phenotype of hemophilia A patients is not only reflected by the actual factor VIII activity level, as there is a large variety in bleeding among patients with similar factor VIII activity.

Currently, patients with severe Hemophilia A are treated with either FVIII containing products or Emicizumab. Initially emicizumab was described for patients who developed inhibitors as inhibitors do not interfere with emicizumab. Despite, bleeding complications still may occur and therefore bypassing therapies are still of great importance. Unfortunately, monitoring treatment with these drugs is a challenge.

Thrombin generation profile may be an additional tool in hemophilia patients to differentiate between bleeding phenotype, to guide prophylactic replacement therapy and adjust bypassing therapy, especially in patients treated with emicizumab. Based on recent studies, thrombin generation as a global hemostasis assay offers an opportunity to assess the hemostatic capacity of patients, and therefore has much potential for monitoring therapy. To facilitate this, a hand-held in vitro diagnostic medical device able to simultaneously measure multiple disease biomarkers with a single drop of blood is currently in development, focusing on simultaneous measurements of Factor VIII activity and Thrombin generation.

Objective: The primary objective of this study is to demonstrate that the version A of the HemA EnzySystem can record thrombin generation within a time frame of 60 min in fresh whole blood samples of patients with hemophilia A treated with Factor VIII Bypassing Agent (FEIBA). As secondary objective, the study results will be validated with a Thrombin Generation Assay (TGA) measured in freshly obtained non frozen plasma.

Study design: This is a cross-sectional observational study. All participants are asked to fill a questionnaire prior to blood collection of four tubes. Blood sample measurements will be conducted within a two-hour time frame using the version A of the HemA EnzySystem and the preparation of plasma using a standard TGA assay. Any remaining blood material will be processed and stored.

Study population: The study population consists of 6 patients treated with FEIBA. In total, at least 24 samples are tested, four for each patient (t=0, 30, 120 and 240 minutes).

ELIGIBILITY:
Inclusion criteria (all of the following)

* Diagnosed with mild (FVIII activity levels 5-40%), moderate (FVIII activity levels 1-5%) or severe hemophilia A (FVIII activity levels <1%)
* With inhibitors
* On prophylactic or on-demand treatment with FEIBA (variation in dosing and duration of therapy use)

Exclusion Criteria:

* use of anticoagulants or platelet antagonists (aspirin or any TAR);
* known allergy to stainless steel;
* a bleeding episode within the last two weeks;
* clinical indication of liver cirrhosis (ultrasonography indication, enlarged spleen, decreased platelet count <100 G/l);
* Signs of inflammation or infection
* Current use of:

NSAIDs; antimicrobial medication; thyroid inhibitors or SSRI's;

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemophilia A patients at the Institute of Hematology and Transfusion Medicine who are on prophylactic or on-demand FEIBA treatment.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2024-03-26 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Time between venipuncture and TGA result | 2 hours
  The primary objective of this study is to demonstrate that the EnzySystem Thrombin Generation assay can record thrombin generation within a time frame of 60 min. Fresh whole blood samples of patients with hemophilia A on prophylactic or on-demand FEIBA treatment are used and tested in a near-patient setting at the Institute of Hematology and Transfusion Medicine (IHiT)

SECONDARY OUTCOMES:
Agreement between TGA obtained with the EnzySystem HemA version A and conventional TGA results | 6 hours
  Outcome of the TGAlum measured with the version A of the HemA EnzySystem will be compared to the reference TGA which is the standard method of testing at the IHiT to determine patients coagulation status. The reference TGA will be evaluated using the Ceveron by Technoclone

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology and Blood Transfusion, Warsaw, Mazowieckie Województwo, Poland

IPD SHARING:
Plan to Share IPD: No